CLINICAL TRIAL: NCT02167321
Title: Adjuvant Chemotherapy With FOLFOX After Total Mesorectal Excision for Locally Advanced Rectal Cancer; an Open-label, Multicenter, Prospective, Randomized Phase 3 Trial
Brief Title: Rectal Cancer, Adjuvant Chemotherapy, FOLFOX(5-fluorouracil/Leucovorin/Oxaliplatin), Total Mesorectal Excision
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Joong Bae Ahn, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0239
Record Dates: First submitted 2014-06-11; First posted 2014-06-19 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Arm A; standard neoadjuvant chemoradiotherapy group
  fluoropyrimidine based concurrent chemoradiotherapy-> TME -> adjuvant chemotherapy (Low risk: fluoropyrimidine-based chemotherapy, High risk: FOLFOX)
  Interventions: Drug: Arm A : standard neoadjuvant chemoradiotherapy group
- Arm B (Experimental): Arm B : adjuvant FOLFOX group
  Total mesorectal excision (TME) --> 12 cycles of FOLFOX every 2 weeks (or Total mesorectal excision (TME) --> Concurrent chemoradiotherapy + 12 cycles of FOLFOX every 2 weeks)
  Interventions: Drug: Arm B : adjuvant FOLFOX group

INTERVENTIONS:
Drug: Arm A : standard neoadjuvant chemoradiotherapy group — radiation : 45Gy±5.4Gy/28Fx/5.5weeks concurrent chemoradiotherapy : 5-FU (400 mg/m2, IV bolus on D1-3, D29-31), leucovorin (20 mg/m2, IV bolus on D1-3, D29-31), preoperative capecitabine : 825 mg/m² p.o. twice daily during XRT, postoperative FL : 5-FU (400 mg/m2, IV bolus)+leucovorin (20m g/m2, IV bolus) on days 1-5 of each 28 day postoperative capecitabine : 1250 mg/m² p.o. twice daily on days 1-14 of each 21 day cycle FOLFOX : oxaliplatin 85 mg/m2, IV over 2 hours on day 1 of each 14 day cycle, leucovorin 200 mg/m2, IV over 2 hours on day 1 of each 14 day cycle, 5-FU 400 mg/m2, IV bolus on day 1 followed by 1200mg/m2 IV over 24 hours on days 1 and 2 of each 14 day cycle
  Other Names: fluoropyrimidine based CCRT -> TME -> adjuvant chemotherapy
  Arms: Arm A
Drug: Arm B : adjuvant FOLFOX group — FOLFOX : oxaliplatin (85 mg/m2, IV over 2 hours on day 1 of each 14 day cycle), leucovorin (200 mg/m2, IV over 2 hours on day 1 of each 14 day cycle), 5-FU (400 mg/m2, IV bolus on day 1 followed by 1200mg/m2 IV over 24 hours on days 1 and 2 of each 14 day cycle) postoperative irradiation(if needed) : 54Gy/30Fx/6weeks
  Other Names: Total mesorectal excision (TME) -> 12 cycles of FOLFOX every 2 weeks; or Total mesorectal excision (TME) -> CCRT + 12 cycles of FOLFOX every 2 weeks
  Arms: Arm B

SUMMARY:
The introduction of total mesorectal excision (TME) and the progress of neoadjuvant chemoradiotherapy has significantly reduced the risk of local recurrence in locally advanced rectal cancer. However, systemic recurrence rate is not being improved and that is considered as the cause of unsatisfactory overall survival of patients with rectal cancer. Relatively higher systemic relapse rate than local recurrence rate is probably due to the insufficient control of systemic micrometastasis during adjuvant chemotherapy. The efficacy of adjuvant combination cytotoxic chemotherapy after surgery in treatment of rectal cancer remains controversial. In addition, preoperative radiotherapy increases surgical complication such as anastomosis site leakage and radiotherapy itself worsen sexual and urinary function and bowel habit which result in aggravation of the quality of life. Furthermore the preoperative chemoradiotherapy upto 3 months not only extends treatment period but increases cost of care. To reduce the possibility of overtreatment, it is needed to confirm that the preoperative chemoradiotherapy is absolutely necessary to locally advanced rectal cancer patients with safe circumferential margin (CRM) resected curatively by standardized TME operation.

In this study, investigators aim to evaluate the efficacy of adjuvant FOLFOX chemotherapy after TME without preoperative chemoradiotherapy in patients with locally advanced rectal cancer having spared CRM are not inferior to that of current standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the rectum below 10 cm from the anal verge
2. Locally advanced rectal cancer (T3N0 or T1-3N+)
3. Age: 19-80 years old.
4. Without evidence of distant metastasis including paraortic lymph node, common & external iliac lymph node metastasis
5. MRI scan confirmed more than 2 mm circumferential margin
6. ECOG(Eastern Cooperative Oncology Group) performance status 0-2
7. preoperative ASA class I-III
8. No prior systemic treatment for rectal cancer (i.e. chemotherapy or immunotherapy)
9. No history of regional radiation treatment in the pelvic cavity
10. Adequate hematologic function: ANC(absolute neutrophil count) ≥ 1.5×109/L，Platelet ≥ 100×109/L, Adequate renal function: Cr ≤ 1.5×ULN or Glomerular filtration rate (Ccr calculated by Cockcroft formula) ≥ 50 ml/min, Adequate hepatic function: ALT(Alanine aminotransferase)/AST(aspartate aminotransferase) ≤ 2.5×ULN, Total bilirubin ≤ 1.5×ULN
11. Patients must be willing and able to comply with the protocol duration of the study
12. Signed informed consent

Exclusion Criteria:

1. Malignancy of the rectum other than adenocarcinoma or adenocarcinoma developed from inflammatory bowel disease
2. Suspicious distant metastasis
3. Patients with peripheral neuropathy ≥ NCI CTC(common terminology criteria) grade 1
4. Uncontrolled and significant cardiovascular disease (i.e. NYHA(New York Heart Association) class III or IV heart failure, myocardial infarction within the past 6 months, uncontrolled angina pectoris)
5. Uncontrolled active infection or serious concomitant systemic disorders incompatible with the study
6. Other co-existing malignancy or malignancy within the past 5 years, with the exception of adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin
7. Patients requiring immunosuppressive treatment who received organ transplantation
8. Uncontrolled epilepsy and psychiatric disease
9. Pregnant or lactating patient
10. Females with a positive or no pregnancy test unless childbearing potential can be otherwise excluded (amenorrheic for at least 2 years,hysterectomy or oophorectomy)
11. Patients receiving a concomitant treatment with drugs interacting with 5-Fluorouracil or oxaliplatin such as flucytosine, phenytoin, or warfarin
12. Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-Fluorouracil or known dihydropyrimidine dehydrogenase (DPD) deficiency.
13. Known hypersensitivity to platinum-based drugs, leucovorin or capecitabine
14. Patients taking sorivudine or brivudine
15. Patients taking tegafur, gimeracil, oteracil potassium complex or stopped the medication within 7days before.
16. Patients who have hereditary disease like as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, etc.
17. Participant in any clinical trial within 4 weeks before initiation of the study
18. Treatment with bevacizumab, cetuximab, oxaliplatin or irinotecan before screening

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-12; Primary Completion 2019-05 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 3 years

SECONDARY OUTCOMES:
Disease free survival (DFS) | 5 years
Overall survival (OS) | 3 years and 5 years
Local recurrence rate | 3 years and 5 years
Systemic recurrence rate | 3 years and 5 years
Total score for function of urination (IPSS) and defecation (Wexner's score) | 1 month and 6 months after surgery
Evaluation for rate of various events after surgery | 14 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JB, Kim HS, Jung I, Shin SJ, Beom SH, Chang JS, Koom WS, Kim TI, Hur H, Min BS, Kim NK, Park S, Jeong SY, Baek JH, Kim SH, Lim JS, Lee KY, Ahn JB. Upfront radical surgery with total mesorectal excision followed by adjuvant FOLFOX chemotherapy for locally advanced rectal cancer (TME-FOLFOX): an open-label, multicenter, phase II randomized controlled trial. Trials. 2020 Apr 7;21(1):320. doi: 10.1186/s13063-020-04266-6. PMID 32264919